CLINICAL TRIAL: NCT03482934
Title: Predictors of Left Ventricular Hypertrophy in Hypertensive Patients in Assiut Governorate
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nardeen Beshay, Principal investigator, Assiut University
Other Study IDs: LVH in HTN
Record Dates: First submitted 2018-01-03; First posted 2018-03-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-01

CONDITIONS: HTN; Hypertrophy, Left Ventricular
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Sphygmomanometers; Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertensive patients
  Interventions: Device: sphygmomanometer; Device: mobilogragh; Diagnostic Test: ECG; Diagnostic Test: Echocardiography

INTERVENTIONS:
Device: sphygmomanometer — device used for measurement of brachial blood pressure
Device: mobilogragh — device used for measurement of central blood pressure
Diagnostic Test: ECG — Electrocardiogram
Diagnostic Test: Echocardiography — Echocardiography

SUMMARY:
To recognize predictors of left ventricular hypertrophy in hypertensive patients in Assiut government & to recognize the prognostic effect of central blood pressure measurement versus office brachial blood pressure measurement.

DETAILED DESCRIPTION:
Many cohort studies have demonstrated that hypertension is a strong risk factor for total mortality and cardiovascular disease (CVD) in both developing and developed countries.

Although brachial blood pressure (BP) mea¬surements have been used for over a century more and more data suggest that measuring of brachial BP has important limitations. First, a few office BP readings may not be representa¬tive of BP during a patient's daily life. Second, brachial BP may differ from systolic BP mea¬sured at the level of the ascending aorta, i.e. central BP, which is responsible for left ventri¬cle afterload and determines blood flow through coronary and brain arteries .

Recent data from the Strong Heart Study confirm earlier results from smaller studies on high-risk patients that central pulse pressure is superior to brachial pulse pressure in the prediction of further cardiovascular events.

The results of the Conduit Artery Function Evaluation (CAFE) study reminded clinicians of the importance of CBP. Those results demonstrated significant differences in CBP (central SBP and PP) between patient groups treated with different antihypertensive regimens even though peripheral BP levels were comparably lowered, and suggested the potential superiority of CBP to cuff brachial BP in cardiovascular prognostic predictive value in hypertensive patients.

Modifiable risk factors for CVD that are common among adults with hypertension include cigarette smoking/tobacco smoke exposure, DM, dyslipidemia (including high levels of low-density lipoprotein cholesterol or hypercholesterolemia, high levels of triglycerides, and low levels of high-density lipoprotein cholesterol), overweight/obesity, physical inactivity/low fitness level, and unhealthy diet .

There are clear examples around the world of ethnic variations in response to drug therapies epitomized by the benefits of thiazide diuretics and calcium channel blockers in lowering BP in blacks and perhaps in older people of all races, whereas blockers of the renin angiotensin system and β-adrenoceptor receptor blockers are just as effective in some other populations.

Urbanization is a factor that profoundly affects BP patterns. In developed countries, hypertension is more common in rural populations than in urban. This pattern is reversed in developing, lower-, and middle-income countries where the first impact of rising rates of hypertension is seen in urban communities.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patient recorded in our outpatient clinic during the last two years will be included retrospectively & new hypertensive patients presenting to our outpatient clinic will be included prospectively for 1 year .

Exclusion Criteria:

* Patient aged less than 18 year old.
* Patients from outside Assiut government .
* Ischemic heart diasease .
* Heart failure .
* Cerebrovascular stroke .
* Diabetes mellitus .
* Patients on regular dialysis .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patient recorded in our outpatient clinic during the last two years will be included retrospectively & new hypertensive patients presenting to our outpatient clinic will be included prospectively for 1 year .
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between brachial blood pressure (measured by sphygmomanometer ) and left ventricular mass index measured by echocardiography to recognize predictors of left ventricular hypertrophy in HTN patients | baseline
Correlation between non invasive central blood pressure (measured by mobilograph ) and left ventricular mass index (measured by echocardiography) to recognize predictors of left ventricular hypertrophy in HTN patients | Base line

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university of medicine, Asyut, Egypt